CLINICAL TRIAL: NCT06290661
Title: Prospective, Multicentre, Randomised Withdrawal Design of a Clinical Trial Evaluating the Safety and Efficacy of a Percutaneous Peripheral Nerve Stimulation System for Patients With Peripheral Neuropathic Pain.
Brief Title: Clinical Trial of the Safety and Efficacy of Peripheral Nerve Stimulation in the Treatment of Peripheral Neuropathic Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Second People's Hospital of GuangDong Province (Other); Xiamen Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHCT-IEC-SOP-016-03-01
Record Dates: First submitted 2024-02-01; First posted 2024-03-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Postherpetic Neuralgia; Peripheral Neuropathic Pain; Trigeminal Neuralgia
Keywords: Peripheral Nerve Stimulation; peripheral neuropathic pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving active electrostimulation after implantation procedure (Experimental): Twenty-eight participants (anticipated) from different 4 hospital in China whose mean VAS scores decreased more than 30% compared with baseline scores after electrode implantation. They will still receive electrostimulation therapy during randomized withdrawal period.
  Interventions: Device: Active electrostimulation
- Participants receiving placebo electrostimulation after implantation procedure (Placebo Comparator): Twenty-eight participants (anticipated) from different 4 hospital in China whose mean VAS scores decreased more than 30% compared with baseline scores after electrode implantation. The electrostimulation of them will be turned off during randomized withdrawal period.
  Interventions: Device: Placebo electrostimulation

INTERVENTIONS:
Device: Active electrostimulation — Maintain the electrical stimulation state, and according to the patient's feeling to set the appropriate stimulation parameter range (pain relief and no obvious numbness and discomfort), the programme will be written into the patient's self-control remote control, by the patient according to their own pain situation for the independent control of the stimulation current.
  Arms: Participants receiving active electrostimulation after implantation procedure
Device: Placebo electrostimulation — No actual electrostimulation
  Arms: Participants receiving placebo electrostimulation after implantation procedure

SUMMARY:
The goal of this clinical trial is to evaluate safety and efficacy of percutaneous peripheral nerve stimulation in patients with peripheral neuropathic pain. The main questions it aims to answer are:

1. The efficacy of percutaneous peripheral nerve stimulation in patients with peripheral neuropathic pain
2. The safety of percutaneous peripheral nerve stimulation in patients with peripheral neuropathic pain Participants are going to undergo procedure that implant peripheral nerve stimulation electrode produced by Jiangsu CED Medtech Co., Ltd. Then the subjects, whose VAS scores decrease more 30% than baseline level, are classified into two groups randomly. One of the group receiving active stimulation called trial group and another receiving placebo stimulation called control group. All subjects are required to make their own subjects' pain diary to record VSA score before and after implantation until at the end of follow-up. Also, participants are asked to report use of analgesic medications, number of awakenings and adverse events.

Researchers will compare pain scores between the two groups to see if peripheral nerve stimulation is effective to patients with peripheral neuropathic pain.

DETAILED DESCRIPTION:
The investigators divide study process into 3 main periods called enrollment/baseline period, treatment period and follow-up period. The treatment period is classified into test period, randomized withdrawal period and observation period further.

1. Enrollment/baseline period This study will be conducted at four clinical trial sites in China with 3 to 6 subjects included in the pretest and the formal trial planned to enroll 56 subjects. All subjects enter screening process after signing the informed consent form (ICF) approved by the ethics committee. Subjects are enrolled who meet inclusion criteria and do not meet any exclusion criteria. Enrolled subjects will undergo vital signs, physical examination, laboratory tests, and visual analogue scale (VAS) scores for pain for at least 4 days, Neuropathic Pain Scale (DN4), and the Short Form Health Survey (SF-36) as part of the screening period assessment prior to electrode implantation.
2. Treatment period 2.1 Implantation of devices Enrolled subjects are implanted with the percutaneous peripheral nerve stimulation system, which was parameterized by the investigator via a programmable controller. Subjects are provided with a "Transcutaneous Peripheral Nerve Stimulation Remote Control Instruction Manual" to guide them in the proper operation and use of the system.

   2.2 Test period Investigators will adjust stimulation parameters and record VAS score under different parameters conditions. The enrolled subjects are provided 1 to 5 stimulation therapy patterns parameterized by investigators after the test.

   Then the subjects receive continuous stimulation with parameterized patterns of 7 (±3) days and VAS scores are be recorded every day of 7 days. Subjects will enter next stage if their VAS scores decrease more than 30% from baseline level or withdraw the trial as reduction less than 30% and devices are removed.

   2.3 Randomized withdrawal period Subject will be classified into random group. One of the group receiving active stimulation called trial group and another receiving placebo stimulation called control group. Both of two groups are performed stimulation in the next 7 days. The subjects of control group will get active stimulation again as the VAS scores back to and maintain 2 days at baseline level. VAS scores will be recorded every day during this period.

   2.4 Observation period The devices are on work until 28th day after the implantation in trial group; stimulators are turned on after randomized withdrawal period until 28th day after the implantation in control group.

   All subjects have electrode leads removed on day 28 of implantation or at early withdrawal.
3. Follow-up period Investigators will begin follow up as the removal of electrode leads or on the day 28 of implantation. Indicators including VAS score will be evaluated and recorded to assess the efficacy and safety of percutaneous peripheral nerve stimulation during follow-up.

ELIGIBILITY:
Inclusion criteria:

* 18 years old and above, male or female
* Diagnosed by trained clinical doctors as postherpetic neuralgia, which is an indication for peripheral nerve stimulation therapy;
* Assess the damage or disease of the peripheral sensory system through the four questions of Douleur Neuropathy before surgery;
* The subject has received conventional treatment but the efficacy is poor, or cannot tolerate the side effects of conventional treatment;
* Visual analogue scale for pain within 24 hours before surgery ≥ 5;
* The subjects are able to understand the purpose of this study, have sufficient compliance with the research treatment, and are willing to sign an informed consent form;

Exclusion criteria:

* Subjects who need to receive both radio frequency modulation and intrathecal drug infusion treatment simultaneously;
* Subjects who are known to have cardiac implants (pacemakers or defibrillators) or other implantable neural stimulators (spinal cord stimulators or deep brain stimulators, etc.);
* Subjects with severe psychological and/or mental disorders and/or non therapeutic drug dependence;
* Subjects expected to undergo MRI examination within 30 days after PNS implantation;
* Expected to be discharged within 48 hours or less;
* Target nerve damage or muscle defects in known pain areas;
* Subjects who are known to be allergic to skin contact materials (tape or adhesive);
* Allergy to anesthetics such as lidocaine;
* Concomitant severe heart disease, liver disease, kidney disease, respiratory system disease, and coagulation dysfunction;
* Pregnant women, lactating women, or women planning to have children within the next three months;
* Subjects who have participated in any other clinical trial, or who may participate in any other trial after enrollment;
* Other situations that the researcher deems unsuitable for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in mean pain visual analogue scale VAS scores between trial and control groups in the randomised withdrawal period | every day from 7 to 14 days after electrode implantation (randomized withdrawal period)
  Researchers will collect visual analogue scale scores of 7 days after the implantation of peripheral nerve stimulation electrode to calculate mean scores of 4 days before randomized withdrawal and evaluate the difference in pain improvement of peripheral nerve stimulation between the two groups (trial and control group) by analyzing the mean change in VAS scores during randomized withdrawal period.
Visual simulation assessment scale collects pain scores after peripheral electrode placement | Every day from 7 to 28 days after electrode implantation, as well as the 14th day after electrode removal
  Researchers collected daily pain scores from the day of peripheral nerve stimulation electrode implantation until removal using the VAS pain scale, as well as pain scores on the 14th day after electrode removal.

SECONDARY OUTCOMES:
Proportion of subjects whose pain relief more than 30% | Every day for 7 days after electrode implantation (test period)
  The VAS scores recorded in pain diary by participants during randomized withdrawal period decreased more 30% than baseline period.
Proportion of subjects of ideal pain state | Every day for 7 days after electrode implantation (test period), every day from 7 to 14 days after electrode implantation (randomized withdrawal period), and every day from 14 to 28 days after electrode implantation (observation period)
  The VAS scores recorded in pain diary by participants during test period, randomized withdrawal period and observation period less than forty millimeters.
Sleep-related assessment after electrostimulation | Every day for 7 days after electrode implantation (test period), every day from 7 to 14 days after electrode implantation (randomized withdrawal period), and every day from 14 to 28 days after electrode implantation (observation period)
  The number of awakenings in sleep diary by participants during test period, randomized withdrawal period and observation period.
Change of life quality after electrostimulation | 4 days before electrode implantation, 7, 14, 21, 28 days after electrode implantation, and 14 days after electrode removal.
  The subjects will be asked to fulfill the Mos 36-item Short Form Health Survey with assistance of clinical physician.
Analgesic medications | Every day from 4 days before electrode implantation to 14 days after electrode removal.
  Participants themselves record the analgesic medications of name, dosage, numbers, routine and duration after peripheral nerve stimulation.
Stability of external assistant devices | Every day from the 1st to 28th day after electrode implantation, as well as the 14th day after electrode removal.
  The stability is assessed with failure rate which defined as number of failures divided by total number of uses.
Questionnaire survey equipment satisfaction | On the first day of electrode implantation and the day of electrode removal (remove the electrode 28 days after surgery).
  A questionnaire survey (0-10 points, 0 points very dissatisfied, 10 points very satisfied) was conducted for each surgeon on the ease of operation of the product and the reasons for dissatisfaction were recorded; a questionnaire survey (0-10 points, 0 points very dissatisfied, 10 points very satisfied) was conducted for each subject on the comfort and ease of use of the equipment and the reasons for dissatisfaction were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mobbs RJ, Nair S, Blum P. Peripheral nerve stimulation for the treatment of chronic pain. J Clin Neurosci. 2007 Mar;14(3):216-21; discussion 222-3. doi: 10.1016/j.jocn.2005.11.007. PMID 17258129
- [Result] Al-Jehani H, Jacques L. Peripheral nerve stimulation for chronic neurogenic pain. Prog Neurol Surg. 2011;24:27-40. doi: 10.1159/000323017. Epub 2011 Mar 21. PMID 21422774
- [Result] Weiner RL, Reed KL. Peripheral neurostimulation for control of intractable occipital neuralgia. Neuromodulation. 1999 Jul;2(3):217-21. doi: 10.1046/j.1525-1403.1999.00217.x. PMID 22151211
- [Result] Slavin KV. Peripheral nerve stimulation for neuropathic pain. Neurotherapeutics. 2008 Jan;5(1):100-6. doi: 10.1016/j.nurt.2007.11.005. PMID 18164488
- [Result] Gilmore C, Ilfeld B, Rosenow J, Li S, Desai M, Hunter C, Rauck R, Kapural L, Nader A, Mak J, Cohen S, Crosby N, Boggs J. Percutaneous peripheral nerve stimulation for the treatment of chronic neuropathic postamputation pain: a multicenter, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2019 Jun;44(6):637-645. doi: 10.1136/rapm-2018-100109. Epub 2019 Apr 5. PMID 30954936